CLINICAL TRIAL: NCT06481241
Title: Efficacy and Safety of Chemotherapy Combined With CAR-T Cells in Newly Diagnosed Adult Patients With Philadelphia Chromosome-Negative B-cell Acute Lymphoblastic Leukemia
Brief Title: Efficacy and Safety of Chemotherapy Combined With CAR-T Cells in Newly Diagnosed Adult Patients With Ph- B-ALL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024020
Record Dates: First submitted 2024-05-24; First posted 2024-07-01 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Philadelphia Chromosome Negative ALL; Acute Lymphoblastic Leukemia, Adult
Keywords: Philadelphia Chromosome Negative Precursor B-Cell Acute Lymphoblastic Leukaemia; CAR-T cell; Venetoclax; Newly Diagnosed
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Immunotherapy, Adoptive; venetoclax; Genes, bcl-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemotherapy and Sequential CAR-T Cells (Experimental): Ph-ALL patients receiving CAR-T cells as consolidation therapy after achieving complete remission (CR) with pediatric-inspired regimen and venetoclax.
  Interventions: Combination Product: CAR-T cells; Drug: Venetoclax

INTERVENTIONS:
Combination Product: CAR-T cells — CAR-T cells as consolidation therapy
Drug: Venetoclax — VEN
  Other Names: Selective inhibitor of B-cell lymphoma 2 (Bcl-2)

SUMMARY:
In recent years, immunotherapy (eg. blinatumomab, inotuzumab ozogamicin, CAR-T cells) has demonstrated a high safety and efficacy profile in relapsed/refractory (R/R）B-ALL. The available data suggest that the advancement of immunotherapy from relapsed/refractory (R/R) field to the frontline setting may be an important approach to increase the depth of remission, which ultimately translates into a survival benefit. In this study, the investigators propose a treatment regimen using CAR-T cell therapy as a consolidation method for Ph- B-ALL patients achieving complete remission (CR) with chemotherapy, aiming to reduce the total cycles of chemotherapy and related toxicities, shorten length of hospitalization, and ultimately improve patients' survival and quality of life.

DETAILED DESCRIPTION:
The CAR-T cells were murine-derived second-generation CD19 CAR-T with a co-stimulation domain of 4-1BB, and the infusion dose was 1×10^6/kg CAR+ cells in a single infusion.

ELIGIBILITY:
Inclusion Criteria:

1. De novo and primary Ph/BCR-ABL1 negative acute lymphoblastic leukemia diagnosed by the bone marrow cytomorphology, immunophenotyping, cytogenetics and molecular biology according to WHO classification
2. Male or female patients aged 18 years or older
3. CD19 expression on blasts
4. Expected survival time greater than 3 months
5. Adequate end organ function as defined by: Total bilirubin ≤ 1.5 x upper limit of normal（ULN）; serum alanine aminotransferase (ALT) and serum aspartate aminotransferase (AST) ≤ 2.5 x ULN or ≤5 x ULN if leukemic involvement of the liver is present; Creatinine ≤ 1.5 x ULN; Serum amylase and lipase ≤ 1.5 x ULN; Alkaline phosphatase ≤ 2.5 x ULN unless considered tumor related; normal electrolytes: Potassium ≥ LLN; Magnesium ≥ LLN; Phosphorus ≥ LLN; Cardiac color Doppler ultrasound ejection fraction ≥ 45%
6. Subject has provided written informed consent prior to any screening procedure

Exclusion Criteria:

1. Burkitt lymphoma/leukemia
2. Acute Leukemia of Ambiguous Lineage
3. Clinical manifestations of active CNS or extramedullary involvement with ALL
4. Female patients who are pregnant or breast feeding
5. Uncontrolled active serious infections that could, in the investigator's opinion, potentially interfere with the completion of treatment
6. Known HIV seropositivity
7. Clinically significant ventricular arrhythmias, unexplained syncope (not vasovagal) or sinus block, history of chronic bradycardia with a high degree of atrioventricular (AV) conduction block (unless a permanent pacemaker is implanted)
8. Any serious psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment
9. Other conditions assessed by the investigators to be inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) | Up to 2 years post-registration
  From CR1 to relapse, death from any cause or last follow-up

SECONDARY OUTCOMES:
MRD-negative complete remission rate measured by flow cytometry. | After induction (4 week)]
  No blasts were detected by flow cytometry when CR criteria were met after induction therapy.
Overall survival (OS) | Up to 5 years post-registration
  From the date of registration to the date of death resulting from any cause.
Event-free survival (EFS) | Up to 5 years post-registration
  From the date of registration to the date of induction failure, relapse, death from any cause, or last follow-up
MRD-negative complete remission rate measured by NGS tracking clonal IG/TR rearrangements | Up to 1 year post-registration
  No clonal IG/TR rearrangements were detected by NGS
Cumulative incidence of relapse (CIR) | Up to 2 years post-registration]
  Calculated with the cumulative incidence method, with death in patients who had a complete hematologic response as a competing risk.
The rate of adverse events | Up to 5 years post-registration
  adverse events during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China